CLINICAL TRIAL: NCT00464139
Title: High Prevalence of Endometriosis in Infertile Women With Normal Ovulation and Normospermic Partners
Brief Title: Prevalence of Endometriosis in a Well Defined Group of Infertile Women
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Christel Meuleman, MD, University Hospitals Leuven
Other Study IDs: EC - 20/03/2007
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Endometriosis; Infertility
Keywords: endometriosis; prevalence; fertility; pain; ultrasound
MeSH Terms: conditions — Endometriosis; Infertility; Pain | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The diagnosis of endometriosis was always confirmed by histological examination of the lesions excised.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The electronic files of all patients who consulted the LUFC since 2003 were searched to select women with at least 1 year of infertility, a regular cycle (variation 21 - 35 days), whose partner had normal sperm according to World Health Organization (WHO) criteria (n = 304).
  After exclusion of 83 (27,3%) patients with a previous laparoscopic diagnosis of endometriosis before referral to our centre, 221 (72,7%) infertile women were included in our study.
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopy
  Other Names: diagnostic laparoscopy; CO2 laser operative laparoscpy

SUMMARY:
At the Leuven University Fertility Centre (LUFC) of the Department of Obstetrics and Gynecology of the University Hospitals Leuven, Belgium, a retrospective epidemiological prevalence study based on an electronic search of patient files was performed to determine the prevalence of histologically proven endometriosis in a subset of infertile women with a regular cycle (variation 21 - 35 days), a partner with normal sperm and no previous surgical diagnosis of endometriosis.

DETAILED DESCRIPTION:
In this study, the electronic files of all patients who consulted the LUFC since 2003 were searched to select women with at least 1 year of infertility, a regular cycle (variation 21 - 35 days), whose partner had normal sperm according to World Health Organization (WHO) criteria (n = 304).

After exclusion of 83 (27,3%) patients with a previous laparoscopic diagnosis of endometriosis before referral to our centre, 221 (72,7%) infertile women were included in our study.

ELIGIBILITY:
Inclusion Criteria:

* all patients who consulted the LUFC since 2003
* with at least 1 year of infertility,
* a regular cycle (variation 21 - 35 days),
* whose partner had normal sperm according to World Health Organization (WHO) criteria.

Exclusion Criteria:

* a previous laparoscopic diagnosis of endometriosis before referral to our centre

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The electronic files of all patients who consulted the LUFC since 2003 were searched to select women with at least 1 year of infertility, a regular cycle (variation 21 - 35 days), whose partner had normal sperm according to World Health Organization (WHO) criteria (n = 304).
  After exclusion of 83 (27,3%) patients with a previous laparoscopic diagnosis of endometriosis before referral to our centre, 221 (72,7%) infertile women were included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The diagnosis of endometriosis was made by the fertility surgeon of the LUFC. | 2003 - 2006

SECONDARY OUTCOMES:
The diagnosis of endometriosis was always confirmed by histological examination. | 2003 - 2006

CONTACTS AND LOCATIONS:
Overall Officials: Christel LC Meuleman, MD, Principal Investigator — University Hospital Gasthuisberg, Leuven, Belgium; Thomas D'Hooghe, MD, PhD, Study Director — University Hospital Gasthuisberg, Leuven, Belgium
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium